CLINICAL TRIAL: NCT05795049
Title: Genetic Carbohydrate Maldigestion as a Model to Study Food Hypersensitivity Mechanism and Guide Personalised Treatment Using a Non-invasive Multiparametric Test (Work Package 1)
Brief Title: Genetic Carbohydrate Maldigestion as a Model to Study Food Hypersensitivity
Acronym: GenMalCarb
Status: Active, not recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: CICbioGUNE (Unknown); Christian-Albrechts-University of Kiel (Unknown); University of Veterinary Medicine Hannover (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20GA093; 288003 (Other: IRAS)
Record Dates: First submitted 2023-01-23; First posted 2023-04-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome (IBS); Sucrase Isomaltase Deficiency
Keywords: nutrigenetics; carbohydrates maldigestion
MeSH Terms: conditions — Irritable Bowel Syndrome; Sucrase-isomaltase deficiency, congenital | interventions — Defecation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and stool sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBS Patient: IBS patient with diarrhoea or alternating bowel habit
  Interventions: Other: Stool and saliva sample collection; Other: Questionnaire completion
- Healthy subject: Participants without IBS
  Interventions: Other: Stool and saliva sample collection; Other: Questionnaire completion

INTERVENTIONS:
Other: Stool and saliva sample collection — Stool and saliva samples collection
Other: Questionnaire completion — Questionnaire on;
  * demographic, ethnicity, IBS subtype, post-infection onset, previous surgeries
  * IBS severity score for adults
  * Hospital Anxiety and Depression scores for adults
  * Somatization score for adults
  * Total glucose and fructose and excess fructose, lactose, sorbitol, mannitol, oligosaccharides (Fructans and GOS) as measured by CNAQ questionnaire for adults and children
  * Quality of Life as measured by the PedsQL™ GI Symptoms Module
  * GI symptoms as measured by the PedsQL™ GI Symptoms Module
  * Anxiety, Depression as measured by the Pediatric PROMIS®

SUMMARY:
Irritable bowel syndrome (IBS) affects one in seven people with gastrointestinal (GI) symptoms. IBS strongly impacts quality of life, is a leading cause of work absenteeism, and consumes 0.5% of the healthcare annual budget. It manifests in women more than men with symptoms including abdominal pain, bloating, constipation (IBS-C), diarrhoea (IBS-D), and mixed presentations (IBS-M) (1). The development of therapeutic options is hampered by the poor understanding of the underlying cause of symptoms.

Many patients find that certain foods (particularly carbohydrates) trigger their symptoms, and avoiding such foods has been shown effective in IBS, like in the low-FODMAP (fermentable oligo-, di-, mono-saccharides and polyols) exclusion diet.

This has suggested that the food-symptom relation may involve malabsorption of carbohydrates due to inefficient digestion. However only a percentage of patients respond to this diet. Recently it has been reported that a subset of IBS carries hypomorphic (defective) gene variant of the sucrase isomaltase (SI), the enzyme that normally digests carbohydrates, sucrose and starch. This carbohydrate maldigestion (the breakdown of complex carbohydrates by a person's small bowel enzymes) is characterized by diarrhoea, abdominal pain and bloating, which are also features of IBS. This possibly occurs via accumulation of undigested carbohydrates in the large bowel, where they cause symptoms due to gas production following bacterial fermentation. Similar mechanisms may be acting at the level of other enzymes involved in the digestion, breakdown and absorption of carbohydrates (carb digestion genes -CDGs). Aim of the study is to study the prevalence of this genetic alteration in a large number of IBS patients as compared to asymptomatic controls.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Patients age between 5 and 70 years of age.
* Patients with IBS-D or IBS-M as defined by the Rome III criteria.
* Previous negative endoscopy with biopsies excluding IBD or microscopic colitis in patients above 50 years old
* Negative relevant additional screening or consultation whenever appropriate
* Ability to conform to the study protocol

Exclusion Criteria for Patients:

* Patients with IBS-C or IBS-U according to Rome III criteria
* Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for participation in the study.
* Patients on opioids
* Patients with concurrent organic gastrointestinal disease (inflammatory bowel disease, celiac disease, cancer), or a major disease such as diabetes, uncontrolled thyroid disease
* Patients with a history of bowel surgery (not appendectomy or cholecystectomy)
* Concurrent major confounding condition, e.g. alcohol or substance abuse in the last 2 years (clinician's judgement).

Inclusion Criteria for healthy controls:

* Between 5 and 70 years of age
* Absence of Rome III IBS criteria

Exclusion Criteria for healthy controls:

* Blood relatives of the participating IBS patient are not allowed to participate.
* Person with any condition which, in the opinion of the investigator, makes them unsuitable for participation in the study.
* Person presenting with a functional or organic GI disorder.
* Person presenting with underlying disease that may involve the GI tract (e.g. Parkinson's disease) or be associated with GI symptoms (e.g. anorexia nervosa, major depression).

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Multicentre study. IBS patients identified through secondary and tertiary care gastroenterological clinics.
  Asymptomatic adult controls recruited at the same site as respective patients or, for instance, from transfusion clinics, blood donor centres, bowel cancer screening as long as data on the absence of symptoms is documented.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
number of IBS-D and IBS-M with of SI and CDG hypomorphic variants as compared to asymptomatic controls | baseline
  the prevalence of SI and CDG hypomorphic variants in IBS-D and IBS-M patients across countries and ethnicities, compared to asymptomatic controls

SECONDARY OUTCOMES:
Difference in age between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - age in years
Difference in gender between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - gender
Difference in ethnicity between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - ethnicity
Difference in IBS subtype between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - number of patients with IBS with diarrhoea (IBS-D) and with mixed bowel habit (IBS-M)
Difference in post-infectious onset between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - number of patients with post-infectious onset
Difference in number of previous abdominal surgery between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - number of patients with IBS with previous abdominal surgery
Difference in symptoms presentations between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - IBS symptoms severity score for adults. This score range between 0 and 500 and a change of at least 50 is considered a clinically relevant change.
Difference in anxiety and depression between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - Hospital Anxiety and Depression score for adults. A score up to 7 for anxiety and or depression is considered Normal; between 8-10 Borderline abnormal (borderline case) and between 11-21 = Abnormal (case)
Difference in somatisation between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - Somatization score for adults. a score of 5, 10, and 15 represent cutpoints for low, medium, and high somatic symptom severity, respectively.
Difference in habitual intake of sugars between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - Total glucose and fructose and excess fructose, lactose, sorbitol, mannitol, oligosaccharides (Fructans and GOS) as measured by CNAQ questionnaire for adults and children
Difference in quality of life between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - Quality of Life as measured by the Pediatric Quality of Life Inventory™ Gastrointestinal Symptoms (PedsQL™ GI Symptoms) Scale. The high.er the PedsQL score, the better the quality of life
Difference in symptoms between patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - GI symptoms using those reported in the Pediatric Quality of Life Inventory™ Gastrointestinal Symptoms Module
Difference in anxiety and depression between paediatric patients carriers and non-carriers of defective (hypomorphic) gene | baseline
  Evaluate whether the below parameters differs between patients carriers and non-carriers of defective (hypomorphic) gene:
  - Anxiety, Depression as measured by the Pediatric Patient-Reported Outcomes Measurement Information System (PROMIS®). This use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric:
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
Difference in in vitro SI enzyme activity in human cells with defective gene as compare with those with normal gene | baseline
  Difference in the intensity of the SI protein bands of immunoprecipitations of monoclonal anti-SI antibodies that recognize different conformations of the SI protein

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ford AC, Lacy BE, Talley NJ. Irritable Bowel Syndrome. N Engl J Med. 2017 Jun 29;376(26):2566-2578. doi: 10.1056/NEJMra1607547. No abstract available. PMID 28657875
- [Background] Shepherd SJ, Lomer MC, Gibson PR. Short-chain carbohydrates and functional gastrointestinal disorders. Am J Gastroenterol. 2013 May;108(5):707-17. doi: 10.1038/ajg.2013.96. Epub 2013 Apr 16. PMID 23588241
- [Background] Eswaran SL, Chey WD, Han-Markey T, Ball S, Jackson K. A Randomized Controlled Trial Comparing the Low FODMAP Diet vs. Modified NICE Guidelines in US Adults with IBS-D. Am J Gastroenterol. 2016 Dec;111(12):1824-1832. doi: 10.1038/ajg.2016.434. Epub 2016 Oct 11. PMID 27725652
- [Background] Ament ME, Perera DR, Esther LJ. Sucrase-isomaltase deficiency-a frequently misdiagnosed disease. J Pediatr. 1973 Nov;83(5):721-7. doi: 10.1016/s0022-3476(73)80362-2. No abstract available. PMID 4742566
- [Background] Chumpitazi BP, Lewis J, Cooper D, D'Amato M, Lim J, Gupta S, Miranda A, Terry N, Mehta D, Scheimann A, O'Gorman M, Tipnis N, Davies Y, Friedlander J, Smith H, Punati J, Khlevner J, Setty M, Di Lorenzo C. Hypomorphic SI genetic variants are associated with childhood chronic loose stools. PLoS One. 2020 May 20;15(5):e0231891. doi: 10.1371/journal.pone.0231891. eCollection 2020. PMID 32433684
- [Background] Henstrom M, Diekmann L, Bonfiglio F, Hadizadeh F, Kuech EM, von Kockritz-Blickwede M, Thingholm LB, Zheng T, Assadi G, Dierks C, Heine M, Philipp U, Distl O, Money ME, Belheouane M, Heinsen FA, Rafter J, Nardone G, Cuomo R, Usai-Satta P, Galeazzi F, Neri M, Walter S, Simren M, Karling P, Ohlsson B, Schmidt PT, Lindberg G, Dlugosz A, Agreus L, Andreasson A, Mayer E, Baines JF, Engstrand L, Portincasa P, Bellini M, Stanghellini V, Barbara G, Chang L, Camilleri M, Franke A, Naim HY, D'Amato M. Functional variants in the sucrase-isomaltase gene associate with increased risk of irritable bowel syndrome. Gut. 2018 Feb;67(2):263-270. doi: 10.1136/gutjnl-2016-312456. Epub 2016 Nov 21. PMID 27872184
- [Background] Garcia-Etxebarria K, Zheng T, Bonfiglio F, Bujanda L, Dlugosz A, Lindberg G, Schmidt PT, Karling P, Ohlsson B, Simren M, Walter S, Nardone G, Cuomo R, Usai-Satta P, Galeazzi F, Neri M, Portincasa P, Bellini M, Barbara G, Jonkers D, Eswaran S, Chey WD, Kashyap P, Chang L, Mayer EA, Wouters MM, Boeckxstaens G, Camilleri M, Franke A, D'Amato M. Increased Prevalence of Rare Sucrase-isomaltase Pathogenic Variants in Irritable Bowel Syndrome Patients. Clin Gastroenterol Hepatol. 2018 Oct;16(10):1673-1676. doi: 10.1016/j.cgh.2018.01.047. Epub 2018 Feb 21. PMID 29408290
- [Background] Thingholm L, Ruhlemann M, Wang J, Hubenthal M, Lieb W, Laudes M, Franke A, D'Amato M. Sucrase-isomaltase 15Phe IBS risk variant in relation to dietary carbohydrates and faecal microbiota composition. Gut. 2019 Jan;68(1):177-178. doi: 10.1136/gutjnl-2017-315841. Epub 2018 Jan 13. No abstract available. PMID 29331942
- [Background] Husein DM, Naim HY. Impaired cell surface expression and digestive function of sucrase-isomaltase gene variants are associated with reduced efficacy of low FODMAPs diet in patients with IBS-D. Gut. 2020 Aug;69(8):1538-1539. doi: 10.1136/gutjnl-2019-319411. Epub 2019 Jul 22. No abstract available. PMID 31331993
- [Background] Zheng T, Eswaran S, Photenhauer AL, Merchant JL, Chey WD, D'Amato M. Reduced efficacy of low FODMAPs diet in patients with IBS-D carrying sucrase-isomaltase (SI) hypomorphic variants. Gut. 2020 Feb;69(2):397-398. doi: 10.1136/gutjnl-2018-318036. Epub 2019 Jan 18. No abstract available. PMID 30658996
- [Background] Spiller RC, Thompson WG. Bowel disorders. Am J Gastroenterol. 2010 Apr;105(4):775-85. doi: 10.1038/ajg.2010.69. No abstract available. PMID 20372130
- [Background] Rasquin A, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006 Apr;130(5):1527-37. doi: 10.1053/j.gastro.2005.08.063. PMID 16678566
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Spiller RC, Humes DJ, Campbell E, Hastings M, Neal KR, Dukes GE, Whorwell PJ. The Patient Health Questionnaire 12 Somatic Symptom scale as a predictor of symptom severity and consulting behaviour in patients with irritable bowel syndrome and symptomatic diverticular disease. Aliment Pharmacol Ther. 2010 Sep;32(6):811-20. doi: 10.1111/j.1365-2036.2010.04402.x. PMID 20629976
- [Background] Varni JW, Bendo CB, Denham J, Shulman RJ, Self MM, Neigut DA, Nurko S, Patel AS, Franciosi JP, Saps M, Verga B, Smith A, Yeckes A, Heinz N, Langseder A, Saeed S, Zacur GM, Pohl JF. PedsQL gastrointestinal symptoms module: feasibility, reliability, and validity. J Pediatr Gastroenterol Nutr. 2014 Sep;59(3):347-55. doi: 10.1097/MPG.0000000000000414. PMID 24806837
- [Background] Irwin DE, Stucky B, Langer MM, Thissen D, Dewitt EM, Lai JS, Varni JW, Yeatts K, DeWalt DA. An item response analysis of the pediatric PROMIS anxiety and depressive symptoms scales. Qual Life Res. 2010 May;19(4):595-607. doi: 10.1007/s11136-010-9619-3. Epub 2010 Mar 7. PMID 20213516
- See also: Sponsor website page — http://www.nuh.nhs.uk/genmalcarb-study/